CLINICAL TRIAL: NCT02624284
Title: tDCS Effects on Resisting Smoking: Dose Ranging Study
Acronym: RDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 823413
Record Dates: First submitted 2015-11-17; First posted 2015-12-08 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Nicotine Addiction
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham dose (Sham Comparator): Participants in this arm will receive the sham transcranial direct current stimulation (tDCS) procedure. During sham tDCS, a 1.0 mA to 2.0 mA current will be delivered for approximately 30 seconds before being extinguished over a course of seconds. Again, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area. Most participants cannot distinguish between real and sham tDCS.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- 1mA dose (Experimental): Participants in this arm will receive the 1mA transcranial direct current stimulation (tDCS) procedure. A neuroConn DC-Stimulator Plus will apply a constant direct current (1.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
  Interventions: Device: transcranial direct current stimulation (tDCS)
- 2 mA dose (Experimental): Participants in this arm will receive the 2 mA transcranial direct current stimulation (tDCS) procedure. A neuroConn DC-Stimulator Plus will apply a constant direct current (2.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Active tDCS: A neuroConn DC-Stimulator Plus will apply a constant direct current (1.0 mA to 2.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
  Sham tDCS: During sham tDCS, a 1.0 mA to 2.0 mA current will be delivered for approximately 30 seconds before being extinguished over a course of seconds. Again, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area. Most participants cannot distinguish between real and sham tDCS.
  Other Names: tDCS, neuroConn DC-Stimulator Plus

SUMMARY:
Behaviors such as tobacco use, unhealthy diet, and sedentary behavior have far-reaching health implications. These modifiable behaviors account for a substantial proportion of deaths from cancer, cardiovascular disease and diabetes, and take a significant economic toll. Yet, many unhealthy behaviors are very resistant to change, despite widespread knowledge of the risks. Although theories of behavior change have been advanced to explain the persistence of these behaviors, few consider the neurobehavioral underpinnings. These approaches also fail to address a fundamental aspect of behavior change - an individual's ability to exert sufficient self-control to overcome temptations for immediate gratification and/or to maintain attention to long-term goals. With advances in the neuroimaging field, the investigators are learning where and how self-control over decisions and behaviors is executed in the brain. This work points to the central role of neural activity in the dorsolateral prefrontal cortices (DLPFC) in self-control processes that contribute to healthy choices. Further, emerging evidence shows that activity in the prefrontal cortices and cognitive control circuits can be modulated using a noninvasive and safe intervention: direct current transcranial stimulation (tDCS). The investigators pilot study, IRB study #820231, demonstrated that a single session of 1mA tDCS increased the ability to resist smoking in a validated smoking lapse paradigm. The current study will use a between-subject design to investigate the dose/response relationship between tDCS (administered at 1mA, 2mA, or sham stimulation for three sessions) and ability to resist smoking.

DETAILED DESCRIPTION:
This trial will use a between-subject single blind design in which participants will be randomized to one of three tDCS dosage groups (1mA, 2mA or sham) and will receive three 20 minute sessions of the same dosage over the course of 1 week before completing a 7 day quit attempt. Eligible participants will complete an Intake Visit (week -1) for final eligibility determination, and complete baseline measures (if eligible). Participants will then be randomly assigned to one of the three dosage groups (1mA, 2mA or sham) and will attend three identical tDCS resist-smoking sessions (study days 1, 3, & 5) during which they will receive 20 minutes of their assigned tDCS dosage and complete cognitive tasks and a resist smoking paradigm. During the resist smoking sessions, participants will receive a session of their assigned dosage of tDCS for 20 minutes while being exposed to in vivo smoking cues (their cigarette pack, cigarettes, an ashtray). Participants will not be informed of their dosage condition. During and after the tDCS session, participants will have the opportunity to smoke in the approved smoking lab. The investigators will measure time to first cigarette and subsequent ad libitum smoking during the resist smoking paradigm. Following Session 3 participants will receive a 20 minute coaching session from a trained smoking cessation counselor to help them prepare for a 7-day quit attempt. During the 7-day quit attempt participants will be asked to attend 4 monitoring visits (study days 6, 8, 10 & 12) to confirm smoking status.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who are between 18 and 60 years of age
2. Report smoking at least 10 cigarettes per day for the past year and have a CO value of > 10ppm at intake
3. Planning to live in the area for at least the next 2 months;
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form;
5. Able to communicate fluently in English (speaking, writing, and reading);
6. Smokers who answer yes on a question regarding motivation to quit smoking.

Exclusion Criteria:

Alcohol/Drugs:

1. History or current diagnosis or treatment for alcohol or drug abuse (as reported during phone screen);
2. Positive breath alcohol concentration test (BrAC >0.01) at any study visit. a. Participants testing positive for breath alcohol with a reading equal to or greater than .08 (the legal driving limit) or who are visibly impaired will be instructed not to drive themselves home after the appointment. If a participant needs to use a phone to call for a safe ride home, an office telephone will be made available to the participant.

Medication:

Current use or recent discontinuation (within the last 14 days at the time of Intake) of:

1. Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix);
2. Anti-psychotic medications;
3. Nicotine replacement therapy (NRT);
4. GABAergic medications;
5. Glutamatergic medications;
6. Any medication that could compromise participant safety as determined by the Principal Investigator and/or Study Physician.

   Daily use of:
7. Opiate-containing medications for chronic pain;
8. Benzodiazepines.

Medical/Neuropsychiatric:

1. Women who are pregnant, planning a pregnancy, and/or breast feeding. All female subjects will complete a urine pregnancy test at the intake visit and preceding all brain stimulation sessions (4 urine pregnancy tests in total);
2. History of epilepsy or a seizure disorder;
3. History of stroke;
4. Self-reported history of brain or spinal tumor;
5. Self-reported history or current diagnosis of psychosis, including schizophrenia, mania, bipolar disorder, major depression (subjects with a history of major depression but in remission for past 6 months are eligible).

tDCS-related:

1. Self-report of metallic objects in the face or head other than dental apparatus (e.g. braces, fillings, and implants);
2. Self-report of pacemakers or implantable cardioverter-defibrillator (ICD).
3. Self-report of any skull fracture or opening.

General Exclusion:

1. Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator;
2. Low or borderline intellectual functioning - determined by a score of less than 90 on the Shipley Institute of Living Scale (SILS) (administered at Intake Visit). The SILS correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test;
3. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Dose: Participants in this arm will receive the sham transcranial direct current stimulation (tDCS) procedure. During sham tDCS, a 1.0 mA to 2.0 mA current will be delivered for approximately 30 seconds before being extinguished over a course of seconds. The anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area.
  Sham tDCS: During sham tDCS, a 1.0 mA to 2.0 mA current will be delivered for approximately 30 seconds before being extinguished over a course of seconds. Again, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area. Most participants cannot distinguish between real and sham tDCS.
- 1mA Dose: Participants in this arm will receive the 1mA transcranial direct current stimulation (tDCS) procedure. A neuroConn DC-Stimulator Plus will apply a constant direct current (1.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
  transcranial direct current stimulation (tDCS): Active tDCS: A neuroConn DC-Stimulator Plus will apply a constant direct current (1.0 mA to 2.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
- 2 mA Dose: Participants in this arm will receive the 2 mA transcranial direct current stimulation (tDCS) procedure. A neuroConn DC-Stimulator Plus will apply a constant direct current (2.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
  transcranial direct current stimulation (tDCS): Active tDCS: A neuroConn DC-Stimulator Plus will apply a constant direct current (1.0 mA to 2.0 mA via 5x7 electrode) to the left dorsal lateral prefrontal cortex. Each participant will receive anodal stimulation for a period of 20 minutes. For anodal stimulation over the left DLPFC, the anodal electrode will be placed over the left F3 and the cathodal electrode over the right supraorbital area (international EEG 10/20 system).
Period: Overall Study
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
Started (Only participants who attended their first session of tDCS are included in this number.) | 49 | 53 | 47
Completed | 35 | 35 | 36
Not Completed | 14 | 18 | 11
Not completed — Withdrawal by Subject | 3 | 6 | 3
Not completed — Protocol Violation | 9 | 10 | 7
Not completed — Revealed exclusionary condition | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose | Total
Number analyzed (Participants) | 35 | 35 | 36 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.2) | 45.6 (9.4) | 45.4 (9.2) | 45.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 10 | 38
  Male | 20 | 22 | 26 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 25 | 28 | 77
  White | 10 | 8 | 7 | 25
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 36 | 106
Nicotine dependence (FTND score) [Mean (Standard Deviation); unit: units on a scale] — The Fagerstrom Test for Nicotine Dependence (FTND) is a validated 6-item measure assessing physical and physiological symptoms of nicotine dependence. The range of scores possible is 0-9; higher scores indicate greater levels of dependence.
  units on a scale | 5.3 (1.5) | 5.1 (1.6) | 5.1 (1.8) | 5.2 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Resisting Smoking - Time to First Cigarette in the Resist Smoking Paradigm
Description: Participant smoking behavior will be assessed during the laboratory session using a validated smoking lapse paradigm. The primary outcome measure is time to first cigarette in minutes.
Time Frame: During laboratory session on day 5, assessed for up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
Number analyzed (Participants) | 35 | 35 | 36
minutes | 60.3 (5.2) | 63.4 (5.4) | 63.2 (4.7)
Statistical Analysis 1: Comparison: Sham Dose vs 1mA Dose vs 2 mA Dose; Test type: Superiority — Analysis: Multiple regression predicting main effects of dose on latency to smoke. Age, sex, race, nicotine dependence, and pre-session craving for negative affect relief (QSU-B Factor 2) were included as covariates; p = 0.94, Regression, Linear

2. Primary Outcome: Resisting Smoking - Number of Cigarettes Smoked in the Resist Smoking Paradigm
Description: Participant smoking behavior will be assessed during the laboratory session using a validated smoking lapse paradigm. The primary outcome measure is number of cigarettes smoked.
Time Frame: During laboratory session on day 5, assessed for up to 2 hours
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
Number analyzed (Participants) | 35 | 35 | 36
cigarettes | 1.6 (0.21) | 1.4 (0.19) | 1.5 (0.18)
Statistical Analysis 1: Comparison: Sham Dose vs 1mA Dose vs 2 mA Dose; Test type: Superiority — Analysis: Multiple regression predicting main effects of dose on number of cigarettes smoked. Age, sex, race, nicotine dependence, and pre-session craving for negative affect relief (QSU-B Factor 2) were included as covariates; p = 0.53, Regression, Linear

3. Secondary Outcome: Urge to Smoke for Negative Affect Relief
Description: The 10-item brief QSU (QSU-B) questionnaire will be used to assess smoking urges. The QSU-B contains 2 subscales (anticipation of reward, relief from negative affect). The QSU-B with a "Right Now" frame of reference will be administered before the smoking resist paradigm. Urge to smoke for negative affect relief (QSU-B Factor 2) has been linked to outcomes for the smoking resist paradigm. The range of possible scores is 4 to 28, with higher scores indicating greater urges.
Time Frame: During laboratory session on day 5, assessed for up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
Number analyzed (Participants) | 35 | 35 | 36
units on a scale | 11.5 (4.9) | 10.8 (6.5) | 8.6 (5.4)

4. Secondary Outcome: Number of Days Abstinent From Cigarettes During Monitored Abstinence Period
Description: Number of days of biochemically verified abstinence during the monitoring period will be recorded.
Time Frame: Assessed during 7-day monitored abstinence period during study days 6 - 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
Number analyzed (Participants) | 35 | 35 | 36
Days | 3.8 (0.43) | 4.1 (0.44) | 3.6 (0.4)
Statistical Analysis 1: Comparison: Sham Dose vs 1mA Dose vs 2 mA Dose; Test type: Superiority — Analysis: Multiple regression predicting main effects of dose on days of abstinence. Age, sex, race and nicotine dependence were included as covariates; p = 0.78, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Sham Dose | 1mA Dose | 2 mA Dose
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/53 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 1/53 | 3/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Dose (N=49) | 1mA Dose (N=53) | 2 mA Dose (N=47)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
high blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bike accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tingling and burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02624284/Prot_SAP_000.pdf